CLINICAL TRIAL: NCT07382947
Title: EXAMINING MENSTRUAL MANAGEMENT AMONG WOMEN OF DIFFERENT GENERATIONS
Brief Title: MENSTRUATİON MANAGEMENT ACCORDİNG TO GENERATİONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, merve yiğit kocamer, DR, Batman University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAU-FTR-MYK-03
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Menstrual Management; Generational Differences; Womens Health; Menstrual Health
Keywords: menstrual management; generational differences; womens health; menstrual health

STUDY DESIGN:
Intervention Model Description: Generation X group Generation Y group Generation Z group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- X generation (Active Comparator): Data will be collected online (Google Forms) on a voluntary basis. At the beginning of the survey, participants will be presented with the purpose of the research, privacy principles, and an informed consent form.
  Interventions: Other: survey data entry
- Y Generation (Active Comparator): Data will be collected online (Google Forms) on a voluntary basis. At the beginning of the survey, participants will be presented with the purpose of the research, privacy principles, and an informed consent form.
  Interventions: Other: survey data entry
- Z Generation (Active Comparator): Data will be collected online (Google Forms) on a voluntary basis. At the beginning of the survey, participants will be presented with the purpose of the research, privacy principles, and an informed consent form.
  Interventions: Other: survey data entry

INTERVENTIONS:
Other: survey data entry — survey data entry

SUMMARY:
The most common symptom that occurs during the menstrual cycle is cramping pain in the lower abdomen. This pain during the menstrual cycle is called dysmenorrhea. It is one of the most common causes of pelvic pain in women. Dysmenorrhea is categorized into two types: primary and secondary. Primary dysmenorrhea manifests as painful cramps during the menstrual period without a pelvic pathology. The pain can radiate to the lower back, pelvis, and upper thigh. Although the etiology of primary dysmenorrhea is not fully known, four main causes have been identified. The etiology of primary dysmenorrhea is endocrine causes, increased prostaglandin levels, increased uterine activity, and psychological causes. Among these factors, increased uterine contractions are thought to be particularly effective in causing the pain. Ischemia in the uterus, which occurs with increased contractions, is among the factors that increase the pain. Primary dysmenorrhea has a prevalence ranging from 45% to 95%. Secondary dysmenorrhea, on the other hand, results from underlying pathological causes such as endometriosis, adenomyosis, uterine fibroids, or pelvic infections. Common symptoms of dysmenorrhea include lower abdominal pain along with headache, numbness, sleep disturbances, depression, vomiting, tender breasts, nausea, diarrhea, and increased urine output.

DETAILED DESCRIPTION:
Research objective/rational: The menstrual cycle (MCC) is a physiological process lasting 23-35 days, consisting of two main phases: follicular (from menstruation to ovulation) and luteal (from ovulation to menstruation), characterized by regular fluctuations in estrogen and progesterone hormones. During the menstrual period, estrogen and progesterone levels are low, while in the follicular phase, estrogen increases and peaks at ovulation; at this time, the increase in FSH and LH triggers ovulation. In the luteal phase, progesterone levels rise and peak in the mid-luteal phase, while a second increase in estrogen levels is observed. When fertilization does not occur, both hormones rapidly decrease in the premenstrual period. Mood changes along with these hormonal fluctuations; negative mood increases during the premenstrual and menstrual periods, while positive mood increases during the ovulation period. These changes can negatively affect women's physical activities, work performance, social relationships, and quality of life. The literature reports that women lose more workdays due to health reasons compared to men, and one of the important reasons for this is symptoms associated with the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Being female
* Being between 18-55 years of age
* Having a menstrual cycle
* Voluntarily agreeing to participate in the study
* Approving the informed consent form

Exclusion Criteria:

* Having a serious chronic or neurological disease
* Using hormonal treatment or birth control method (within the last 6 months)
* Being pregnant or in menopause
* Having an incomplete or incorrectly completed questionnaire

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 1200 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Menstruation Symptom Scale (MSQ) | 15 minute
  Developed by Chesney and Tasto in 1975, the MSQ was adapted into Turkish by Güvenç et al. in 2014.
  The scale is a five-point Likert-type scale consisting of 22 items. Participants rate menstruation-related symptoms on a scale of 1 (never) to 5 (always).
  The scale is divided into three sub-dimensions: 'Negative Effects/Somatic Complaints', 'Menstrual Pain Symptoms', and 'Coping Mechanisms'.
  The MSQ score is calculated from the average scores of the items, and a higher score indicates an increase in the severity of symptoms.
Attitude Toward Menstrution Scale: | 15 minute
  Attitude Toward Menstruation Scale: The Turkish validity and reliability study of the scale developed by Brooks-Gunn and Ruble in 1980 was conducted by Kulakaç et al. in 2008. The adapted version of the scale, which is originally a 7-point Likert type, is a 5-point Likert type with a scoring range of 1-5 (1-Strongly disagree, 5-Strongly agree). The scale, which contains a total of 31 items, has 5 sub-dimensions: "Menstruation as a debilitating event" (7 items), "Menstruation as a disturbing event" (5 items), "Menstruation as a natural event" (5 items), "Noticing/sensing changes before and during menstruation" (8 items), "Denial of the effects of menstruation" (6 items). A high average score on the sub-dimensions or the entire scale indicates a "positive" attitude towards menstruation.
WaLIDD (Working ability, Location, Intensity, Days of pain, Dysmenorrhea) Scale: | 5 minute
  It was first developed by Teherán et al. (2013) and is designed to assess the severity, duration, location, and impact on daily life of dysmenorrhea (menstrual pain) in women.
  The Turkish adaptation of the scale was carried out by H. Arıkan and E. Erol and published in 2025.
Visual Analog Scale (VAS): | 1 minute
  The Visual Analog Scale (VAS) was used to subjectively determine the pain of the individuals participating in the study.
  Participants will be asked to indicate the intensity of their pain on a 0-10 cm scale.
  1-3 cm will be considered mild, 4-7 cm moderate, and 8-10 cm severe tension.
Turkish Health Literacy Scale (TSOY-32): | 5 minute
  It is a scale developed to measure individuals' ability to find, understand, evaluate, and use health information. It was adapted to the Turkish society by Abacıgil, Harlak, and Okyay (2016), based on the European Health Literacy Scale (HLS-EU-Q47). The scale, consisting of a total of 32 items, evaluates in three main areas: health services, disease prevention, and health promotion. In the validity and reliability analyses, Cronbach's α value was found to be 0.89.
Step Count: | 1 minute
  The WHO defines mobile health as the support of medical and public health applications by mobile devices such as mobile phones, patient monitoring devices, and other wireless devices.
  Mobile phones are the most commonly used devices in the implementation of mobile health (WHO, 2011). Many studies have reported that pedometers installed on smartphones provide accurate step counting at different walking speeds and with different carrying methods (Funk et al., 2018; Thomson et al., 2019). A-B Participants' physical activity levels were monitored for 7 days through the Google Fit application installed on smartphones. The application automatically records the daily step count, distance covered, and estimated energy expenditure using the device's accelerometer sensor. Participants were asked to keep their phones on them throughout the day and to keep the application open in the background. The average daily step count obtained at the end of 7 days was evaluated as an indicator o
Pittsburgh Sleep Quality Index (PSQI): | 5 minute
  Developed by Buysse and colleagues in 1989, the PSQI is a self-report questionnaire that assesses sleep quality and disturbances over the past month.
  A validity and reliability study conducted in Turkey by Ağargün and colleagues proved that the PSQI is consistent and valid in Turkish society. This scale, consisting of 24 questions, comprises 19 questions based on the individual's self-assessment and 5 questions answered by a spouse or roommate. Each question is scored between 0 and 3 to calculate the total score. A score of five or higher is generally considered poor sleep quality.
Short Form-12 (SF-12): | 5 minute
  Participants' health-related quality of life was assessed using the Short Form-12 (SF-12) scale.
  SF-12 is a short questionnaire consisting of two sub-dimensions, physical and mental health, measuring participants' general health status and quality of life. The physical component score (Physical Component Summary, PCS) and the mental component score (Mental Component Summary, MCS) were calculated separately, with higher scores indicating better quality of life. The Turkish validity and reliability of the scale were established by Demiral et al. (2006).

CONTACTS AND LOCATIONS:
Overall Officials: merve yiğit kocamer, lecturer, Principal Investigator — Batman University
Locations (1):
- Batman Center, Batman, Gültepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No